CLINICAL TRIAL: NCT04268940
Title: Thrombo-Elastography Guided Management of ECMO
Acronym: TEGMO
Status: Completed | Type: Observational
Sponsor: Damian Ratano (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Sponsor-Investigator, Damian Ratano, Principal investigator, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Other Study IDs: 19-5121
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Extracorporeal Circulation of Blood; Thrombocytopenia
Keywords: Unfractionated heparin; Extracorporeal Membrane Oxygenation (ECMO); Thromboelastography; Anticoagulation monitoring; aPTT; Anti-factor Xa; Point-of-care
MeSH Terms: conditions — Thrombocytopenia | interventions — Thrombelastography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Thromboelastography — Thromboelastography (TEG 6s, global hemostasis cartridge) will be performed before ECMO insertion and at different time-points during the course of ECMO. In parallel a full coagulation work-up (aPTT, prothrombin time [PT], anti-Xa, activated clotting time[ACT], platelets count, d-dimers, von Willebrand panel and fibrinogen) will be measured simultaneously with each TEG.

SUMMARY:
Anticoagulation and coagulation management during ECMO is a challenge. Bleeding and clotting are major sources of morbidity and mortality. The currently used strategies are of poor evidence. This observational study wants to evaluate the use of automated thromboelastography (TEG 6s) to guide the management of coagulation and anticoagulation in patients supported by ECMO

DETAILED DESCRIPTION:
ECMO induces both a risk of clotting and bleeding. Therapeutic anticoagulation is recommended during ECMO. While preventing clotting, anticoagulation triggers a higher risk of bleeding. However, anticoagulation does not completely avoid clotting due to complex interactions between the circuit, the patients' blood and the anticoagulant. Unfractionated heparin (UFH) is the most commonly used anticoagulant and requires monitoring. No clear recommendation exists. The activated partial thromboplastin time (aPTT) as well as the anti-factor Xa activity (anti-Xa) are plasma-based tests used to monitor UFH. The evidence for their use is poor and they do no correlate well. Moreover, these two tests do not take into account all the elements of blood and do not reflect the entire coagulation process.

Thromboelastography is a whole-blood point-of-care test that describes each phases of the clotting process from the activation of coagulation factors to the later lysis to the thrombus. TEG is also sensitive to UFH and can be used to quantify its effect. The use of heparinase during TEG also permits to evaluate the coagulation process during the use of heparin. This could give an important understanding of the effect of the ECMO itself on the circuit and help to develop a strategy to prevent bleeding and clotting as well as monitor heparin treatment.

The hypothesis for this study is that the use of thromboelastography will identify situations with high risk of bleeding and allow interventions to reduce hemorrhagic events and blood products transfusions. It is also hypothesized that the monitoring of unfractionated heparin (UFH) with TEG is feasible and could lead to the use of less UFH during the course of ECMO.

The objectives of this study are 1) to determine and calibrate the TEG R-time values corresponding to aPTT therapeutic range for patients under therapeutic UFH during ECMO course, 2) to determine the level of correlation of TEG parameters with other anticoagulation tests [Prothrombin Time (PT), anti-Xa, activated clotting time (ACT)], fibrinogen level, platelets count and d-dimers, 3) to determine the TEG values that are associated with the administration of blood-derived coagulation products in clinical practice 4) to identify TEG cutoff points that are associated with an increased risk of bleeding/clotting in ECMO patients 5) use these observational data to develop a TEG-based algorithm for anticoagulation management and blood products replacement that could be tested in a future study.

This study will you the last version of TEG, TEG-6s which is a fully automated point-of-care device.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients admitted in Toronto General Hospital Medical Surgical ICU (MSICU) supported with ECMO. Patients cannulated before admission (ECMO retrieval) can also be included

Exclusion Criteria:

* Refusal of consent, unavailability or impossibility to process blood samples before ECMO cannulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients suffering from cardiorespiratory failure and needing Extracorporeal Membrane Oxygenation
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-06-04 (Actual)

PRIMARY OUTCOMES:
Correlation between TEG (R-time K-TEG) and aPTT | 0-10 days
Correlation of TEG parameters with "classical" coagulation tests | 0-10 days
Ability of TEG data to identify patients at higher risk of bleeding (or clotting) during the course of ECMO | 0-10 days

CONTACTS AND LOCATIONS:
Overall Officials: Damian Ratano, MD, Principal Investigator — University Health Network, Toronto; Eddy Fan, MD, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sauer CM, Yuh DD, Bonde P. Extracorporeal membrane oxygenation use has increased by 433% in adults in the United States from 2006 to 2011. ASAIO J. 2015 Jan-Feb;61(1):31-6. doi: 10.1097/MAT.0000000000000160. PMID 25303799
- [Background] Gorbet MB, Sefton MV. Biomaterial-associated thrombosis: roles of coagulation factors, complement, platelets and leukocytes. Biomaterials. 2004 Nov;25(26):5681-703. doi: 10.1016/j.biomaterials.2004.01.023. PMID 15147815
- [Background] Annich GM. Extracorporeal life support: the precarious balance of hemostasis. J Thromb Haemost. 2015 Jun;13 Suppl 1:S336-42. doi: 10.1111/jth.12963. PMID 26149045
- [Background] Zangrillo A, Landoni G, Biondi-Zoccai G, Greco M, Greco T, Frati G, Patroniti N, Antonelli M, Pesenti A, Pappalardo F. A meta-analysis of complications and mortality of extracorporeal membrane oxygenation. Crit Care Resusc. 2013 Sep;15(3):172-8. PMID 23944202
- [Background] Youngs RP, Gatland D, Brookes J. Swallowed radiolucent dental prostheses: risk of extraluminal oesophageal perforation. J Laryngol Otol. 1988 Jan;102(1):71-3. doi: 10.1017/s0022215100104037. No abstract available. PMID 3278070
- [Background] Shimizu M, Morito S, Kawamura Y. [Phlebography of several skin diseases likely to be associated with circulatory disorders of the lower extremity, varicose syndromes and Bazin's disease]. Acta Dermatol Kyoto Engl Ed. 1968 Aug;63(3):259-76. No abstract available. Japanese. PMID 5756960
- [Background] Ratano D, Alberio L, Delodder F, Faouzi M, Berger MM. Agreement between activated partial thromboplastin time and anti-Xa activity in critically ill patients receiving therapeutic unfractionated heparin. Thromb Res. 2019 Mar;175:53-58. doi: 10.1016/j.thromres.2019.01.002. Epub 2019 Jan 7. PMID 30708169
- [Background] Basu D, Gallus A, Hirsh J, Cade J. A prospective study of the value of monitoring heparin treatment with the activated partial thromboplastin time. N Engl J Med. 1972 Aug 17;287(7):324-7. doi: 10.1056/NEJM197208172870703. No abstract available. PMID 5041701
- [Background] Levine MN, Hirsh J, Gent M, Turpie AG, Cruickshank M, Weitz J, Anderson D, Johnson M. A randomized trial comparing activated thromboplastin time with heparin assay in patients with acute venous thromboembolism requiring large daily doses of heparin. Arch Intern Med. 1994 Jan 10;154(1):49-56. PMID 8267489
- [Background] Atallah S, Liebl M, Fitousis K, Bostan F, Masud F. Evaluation of the activated clotting time and activated partial thromboplastin time for the monitoring of heparin in adult extracorporeal membrane oxygenation patients. Perfusion. 2014 Sep;29(5):456-61. doi: 10.1177/0267659114524264. Epub 2014 Feb 25. PMID 24570077
- [Background] Panigada M, E Iapichino G, Brioni M, Panarello G, Protti A, Grasselli G, Occhipinti G, Novembrino C, Consonni D, Arcadipane A, Gattinoni L, Pesenti A. Thromboelastography-based anticoagulation management during extracorporeal membrane oxygenation: a safety and feasibility pilot study. Ann Intensive Care. 2018 Jan 16;8(1):7. doi: 10.1186/s13613-017-0352-8. PMID 29340875
- [Background] Henderson N, Sullivan JE, Myers J, Wells T, Calhoun A, Berkenbosch J, Tzanetos DT. Use of Thromboelastography to Predict Thrombotic Complications in Pediatric and Neonatal Extracorporeal Membranous Oxygenation. J Extra Corpor Technol. 2018 Sep;50(3):149-154. PMID 30250340
- [Background] Riley JB, Schears GJ, Nuttall GA, Oliver WC Jr, Ereth MH, Dearani JA. Coagulation Parameter Thresholds Associated with Non-Bleeding in the Eighth Hour of Adult Cardiac Surgical Post-Cardiotomy Extracorporeal Membrane Oxygenation. J Extra Corpor Technol. 2016 Jun;48(2):71-8. PMID 27578897
- [Background] Gurbel PA, Bliden KP, Tantry US, Monroe AL, Muresan AA, Brunner NE, Lopez-Espina CG, Delmenico PR, Cohen E, Raviv G, Haugen DL, Ereth MH. First report of the point-of-care TEG: A technical validation study of the TEG-6S system. Platelets. 2016 Nov;27(7):642-649. doi: 10.3109/09537104.2016.1153617. Epub 2016 Apr 11. PMID 27809712
- [Background] Delmas C, Jacquemin A, Vardon-Bounes F, Georges B, Guerrero F, Hernandez N, Marcheix B, Seguin T, Minville V, Conil JM, Silva S. Anticoagulation Monitoring Under ECMO Support: A Comparative Study Between the Activated Coagulation Time and the Anti-Xa Activity Assay. J Intensive Care Med. 2020 Jul;35(7):679-686. doi: 10.1177/0885066618776937. Epub 2018 May 16. PMID 29768983
- See also: Extracorporeal life support organisation (ELSO) anticoagulation guidelines — https://www.elso.org/Portals/0/Files/elsoanticoagulationguideline8-2014-table-contents.pdf
- See also: TEG 6s description — https://teg.haemonetics.com/en-gb/teg-6s-hemostasis-analyzer